CLINICAL TRIAL: NCT00801879
Title: Intranasal Mupirocin to Eliminate Carriage of Staphylococcus Aureus in HIV Infection
Brief Title: Mupirocin Ointment to Eliminate Nasal Carriage of Staphylococcus Aureus in HIV Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: GlaxoSmithKline (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Franklin D. Lowy, Professor of Medicine and Pathology at the New York-Presbyterian Hospital at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAB0129; K08AI072043 (NIH)
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Staphylococcus Aureus; HIV Infections
Keywords: mupirocin; Staphylococcus aureus; colonization; infection; HIV
MeSH Terms: conditions — Staphylococcal Infections; HIV Infections; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mupirocin ointment (Active Comparator): 0.25g mupirocin calcium ointment, 2% in each nostril twice daily for 5 days (repeated monthly for up to 8 months)
  Interventions: Drug: Mupirocin calcium ointment, 2%
- Placebo ointment (Placebo Comparator): 0.25g in each nostril twice daily for 5 days (repeated monthly for up to 8 months)
  Interventions: Drug: Placebo ointment

INTERVENTIONS:
Drug: Mupirocin calcium ointment, 2% — 0.25 g in each nostril twice daily for 5 days (given monthly for up to 8 months)
  Other Names: Bactroban Nasal 2%
  Arms: Mupirocin ointment
Drug: Placebo ointment — Placebo ointment 0.25g in each nostril twice daily for 5 days (repeated monthly for up to 8 months)
  Arms: Placebo ointment

SUMMARY:
Staphylococcus aureus is a bacteria that causes serious, often life threatening infections including pneumonia, wound, and bloodstream infections. Persons with AIDS are at high risk for S. aureus infections. They are also at high risk for nasal carriage of S. aureus. In fact, nasal carriage is a known risk factor for subsequent S. aureus infection. Topical mupirocin, an antibiotic when applied to the anterior nares, is a safe, effective way to eliminate S. aureus colonization. Some studies have shown that mupirocin can also decrease the risk of S. aureus infection, but many of those studies utilized historical controls and none were rigorously tested among AIDS patients over an extended period of time.

The main purpose of this randomized, double-blinded, placebo controlled study is to determine if mupirocin can eliminate S. aureus nasal colonization in residents at PSI (inpatient, drug rehabilitation facility for AIDS patients in the Bronx.) PSI residents currently have a high incidence of S. aureus nasal colonization and infection. Nasal cultures followed by twice daily application of mupirocin vs. placebo for five days will be performed on a monthly basis for 8 months. the study will examine whether mupirocin decreases the incidence of S. aureus infections and prevents S. aureus nasal colonization. The study is important because it may show that mupirocin is an effective way to eliminate nasal colonization and prevent S. aureus infections in AIDS patients, among those at highest risk for serious S. aureus infection.

Hypothesis: Monthly application of mupirocin will reduce nasal colonization with S.aureus

DETAILED DESCRIPTION:
This was a randomized double-blinded placebo controlled trial. Subjects were treated with intranasal mupirocin or placebo on a monthly basis and tested for nasal colonization a month after each treatment. This was performed up to 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Resident at Project Samaritan Inc. (PSI)

Exclusion Criteria:

* Past hypersensitivity to mupirocin or glycerol
* Pregnancy
* Lactation
* Expected discharge from PSI in the following month
* Treatment with intranasal mupirocin within the preceding two months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-09; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Nasal colonization with Staphylococcus aureus | monthly assessment of colonization (~1 month after each treatment)

SECONDARY OUTCOMES:
Infection with Staphylococcus aureus | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Rachel J Gordon, MD, MPH, Study Director — Columbia University; Franklin D Lowy, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - Project Samaritan Inc., The Bronx, New York

REFERENCES:
- [Result] Gordon RJ, Chez N, Jia H, Zeller B, Sobieszczyk M, Brennan C, Hisert KB, Lee MH, Vavagiakis P, Lowy FD. The NOSE study (nasal ointment for Staphylococcus aureus eradication): a randomized controlled trial of monthly mupirocin in HIV-infected individuals. J Acquir Immune Defic Syndr. 2010 Dec;55(4):466-72. doi: 10.1097/QAI.0b013e3181ec2a68. PMID 20686410